CLINICAL TRIAL: NCT04903093
Title: A PHASE 1, RANDOMIZED, CROSSOVER STUDY TO EVALUATE RELATIVE BIOAVAILABILITY OF ABROCITINIB ORAL SUSPENSION AND EFFECT OF AN ACID-REDUCING AGENT ON THE BIOAVAILABILITY OF ABROCITINIB COMMERCIAL TABLET AND TO ASSESS THE TASTE OF ABROCITINIB ORAL FORMULATIONS IN HEALTHY ADULT PARTICIPANTS AGED 18 TO 55 YEARS OF AGE.
Brief Title: A Study Evaluating Relative Bioavailability of an Oral Suspension of Abrocitinib and Effect of an Acid Reducing Agent on the Bioavailability of Abrocitinib and Assessing the Taste of Abrocitinib Oral Formulations.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7451061
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: Abrocitinib; Atopic Dermatitis; Healthy Volunteers; Relative Bioavailability; Taste Assessment
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib; Famotidine

STUDY DESIGN:
Masking Description: Part A: open label / Part B: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Part A: Abrocitinib Tablet (Experimental)
  Interventions: Drug: Abrocitinib tablet
- Part A: Abrocitinib Suspension F1 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F1
- Part A: Abrocitinib Tablet + Famotidine (Experimental)
  Interventions: Drug: Famotidine
- Part B: Abrocitinib Suspension F1 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F1
- Part B: Abrocitinib Suspension F2 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F2
- Part B: Abrocitinib Suspension F3 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F3
- Part B: Abrocitinib Suspension F4 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F4
- Part B: Abrocitinib Suspension F5 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F5
- Part B: Abrocitinib Suspension F6 (Experimental)
  Interventions: Drug: Abrocitinib Suspension F6
- Part B: Abrocitinib Suspension F1 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F1; Drug: Famotidine
- Part B: Abrocitinib Suspension F2 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F2; Drug: Famotidine
- Part B: Abrocitinib Suspension F3 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F3; Drug: Famotidine
- Part B: Abrocitinib Suspension F4 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F4; Drug: Famotidine
- Part B: Abrocitinib Suspension F5 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F5; Drug: Famotidine
- Part B: Abrocitinib Suspension F6 + Famotidine (Experimental)
  Interventions: Drug: Abrocitinib Suspension F6; Drug: Famotidine

INTERVENTIONS:
Drug: Abrocitinib tablet — Single dose of abrocitinib 200 mg tablet will be administered after an overnight fast of at least 10 hours.
  Arms: Part A: Abrocitinib Tablet
Drug: Abrocitinib Suspension F1 — Single dose of abrocitinib 200 mg oral suspension formulation 1 will be administered after an overnight fast of at least 10 hours.
  Arms: Part A: Abrocitinib Suspension F1; Part B: Abrocitinib Suspension F1; Part B: Abrocitinib Suspension F1 + Famotidine
Drug: Abrocitinib Suspension F2 — Single dose of abrocitinib 200 mg oral suspension formulation 2 will be administered after an overnight fast of at least 10 hours.
  Arms: Part B: Abrocitinib Suspension F2; Part B: Abrocitinib Suspension F2 + Famotidine
Drug: Abrocitinib Suspension F3 — Single dose of abrocitinib 200 mg oral suspension formulation 3 will be administered after an overnight fast of at least 10 hours.
  Arms: Part B: Abrocitinib Suspension F3; Part B: Abrocitinib Suspension F3 + Famotidine
Drug: Abrocitinib Suspension F4 — Single dose of abrocitinib 200 mg oral suspension formulation 4 will be administered after an overnight fast of at least 10 hours.
  Arms: Part B: Abrocitinib Suspension F4; Part B: Abrocitinib Suspension F4 + Famotidine
Drug: Abrocitinib Suspension F5 — Single dose of abrocitinib 200 mg oral suspension formulation 5 will be administered after an overnight fast of at least 10 hours.
  Arms: Part B: Abrocitinib Suspension F5; Part B: Abrocitinib Suspension F5 + Famotidine
Drug: Abrocitinib Suspension F6 — Single dose of abrocitinib 200 mg oral suspension formulation 6 will be administered after an overnight fast of at least 10 hours.
  Arms: Part B: Abrocitinib Suspension F6; Part B: Abrocitinib Suspension F6 + Famotidine
Drug: Famotidine — Single dose of famotidine 40 mg tablet administered 2 hours prior to abrocitinib formulations under fasted conditions.
  Arms: Part A: Abrocitinib Tablet + Famotidine; Part B: Abrocitinib Suspension F1 + Famotidine; Part B: Abrocitinib Suspension F2 + Famotidine; Part B: Abrocitinib Suspension F3 + Famotidine; Part B: Abrocitinib Suspension F4 + Famotidine; Part B: Abrocitinib Suspension F5 + Famotidine; Part B: Abrocitinib Suspension F6 + Famotidine

SUMMARY:
This study consists of 2 parts: Part A is to estimate the relative bioavailability of a single 200 mg dose of abrocitinib oral suspension (Test formulation) compared to the commercial abrocitinib tablet (200 mg) (Reference formulation). The effect of an acid-reducing agent on the pharmacokinetics of abrocitinib and its metabolites will also be evaluated by administering abrocitinib 200 mg commercial tablet with or without famotidine 40 mg, as an acid-reducing agent. Part B is to assess the taste and palatability of six different abrocitinib oral suspension formulations. Additionally, the safety and tolerability of abrocitinib tablet (in Part A) and abrocitinib oral suspension formulations (in Part B) will be assessed when given with or without famotidine 40 mg once daily.

DETAILED DESCRIPTION:
This is a Phase 1 randomized study in healthy participants to estimate the relative bioavailability of abrocitinib oral suspension (Test formulation) compared to commercial abrocitinib tablet (Reference formulation) under fasted condition. The effect of an acid-reducing agent on the pharmacokinetics of the commercial tablet formulation will be evaluated by administering abrocitinib 200 mg commercial tablet with famotidine 40 mg, as an acid-reducing agent. Assessment of taste and palatability of six different abrocitinib suspension formulations will also be performed. This study consists of 2 parts, as listed below:

Part A

Part A of the study will be an open label, randomized, single dose, crossover, 3-treatment, 6 sequence, 3-period design in healthy male and/or female adult participants (18-55 years). Healthy participants will be screened within 28 days prior to the first administration of the study intervention to confirm that they meet the participant selection criteria for the study. Eligible participants will be admitted to the CRU on Day -1 and will be confined in the CRU until discharge, on Day 2 of Period 9 in Part B, after completing both Parts A and B of the study. In Part A, participants will be randomized to receive one of the following: a single 200 mg dose of abrocitinib commercial tablet (Treatment A), a single 200 mg dose of abrocitinib oral suspension formulation 1 (Treatment B), or famotidine (40 mg) administered 120 minutes before a single 200 mg dose of abrocitinib commercial tablet (Treatment C). All participants will be fasting for at least 10 hours before taking abrocitinib.

Part B

Part B will be a single-blind, randomized, 6-period, crossover study in healthy male and/or female adult participants (18-55 years). For any new healthy participants joining Part B only, screening will be performed within 28 days prior to the first administration of the study intervention to confirm that they meet the participant selection criteria for the study. New participants enrolled in Part B only will be admitted to the CRU on Day -1 and will be confined in the CRU until discharge, which is Day 2 of Period 9. On Day 1 of each treatment period under fasted conditions, participants will receive a famotidine tablet (40 mg with 240 mL of room temperature water) administered 120 minutes before a single 200 mg dose of abrocitinib oral suspensions (Formulations 1 to 6) or administered a single 200 mg dose of abrocitinib oral suspension alone (Formulations 1 to 6), after a fast of at least 10 hours before abrocitinib administration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination, laboratory tests, and cardiovascular tests.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus infection; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C virus antibody (HCVAb).
* Other acute or chronic medical or psychiatric condition including recent (within the past year).

Evidence or history of clinically significant dermatological condition (eg, atopic dermatitis or psoriasis) or visible rash present during physical examination.

* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
* A positive urine drug test.
* Selected laboratory abnormalities.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* History of tuberculosis (TB) (active or latent).
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline.
* Pregnant female participants; breastfeeding female participants; female participants of childbearing potential who are unwilling or unable to use an acceptable method of contraception.
* History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A was a crossover, 3-treatment, 6-sequence, 3-periods design. With completion of Part A of the study, participants entered Part B, which included 6 periods with 6 sequences.
  Thus, participants who completed Part A and then Part B were combined. Enrolled participants, including 18 participants who completed both Parts A and B and 1 participant who withdrew by the participant, are presented in the Participant Flow.
Groups:
- Treatment A-> B-> C-> D-> E-> F-> G-> H-> I; Treatment A-> C-> B-> L-> M-> N-> B-> J-> K; Treatment B-> A-> C-> K-> L-> M-> N-> B-> J; Treatment B-> C-> A-> I-> D-> E-> F-> G-> H; Treatment C-> A-> B-> H-> I-> D-> E-> F-> G; Treatment C-> B-> A-> J-> K-> L-> M-> N-> B: Part A of the study included administration of treatments A - C. A=a single dose of abrocitinib 200 mg commercial tablet; B=a single dose of abrocitinib 200 mg oral suspension formulation 1, C=famotidine (40 mg) administered 120 minutes before a single dose of 200 mg abrocitinib commercial tablet.
  Part B of the study included administration of treatments D - I, famotidine 40 mg tablet + abrocitinib 200 mg oral suspension formulation X (X=1-6), and treatments B, J - N, abrocitinib 200 mg oral suspension formulation X (X=1-6) only.
  All were under fasted state on Day 1 of each period.
Period: Overall Study
Arm/Group | Treatment A-> B-> C-> D-> E-> F-> G-> H-> I | Treatment A-> C-> B-> L-> M-> N-> B-> J-> K | Treatment B-> A-> C-> K-> L-> M-> N-> B-> J | Treatment B-> C-> A-> I-> D-> E-> F-> G-> H | Treatment C-> A-> B-> H-> I-> D-> E-> F-> G | Treatment C-> B-> A-> J-> K-> L-> M-> N-> B
Started | 3 | 3 | 3 | 4 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a phase 1, randomized, crossover designed relative bioavailability (rBA) study conducted in healthy adult participants, including 2 parts to investigate the rBA (part A), and taste and palatability (part B) of different formulations. Participants were all healthy adults and were randomized into the study, and may or may not participate both parts of the study. Thus baseline characteristics of participants were combined.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A-> B-> C-> D-> E-> F-> G-> H-> I | Treatment A-> C-> B-> L-> M-> N-> B-> J-> K | Treatment B-> A-> C-> K-> L-> M-> N-> B-> J | Treatment B-> C-> A-> I-> D-> E-> F-> G-> H | Treatment C-> A-> B-> H-> I-> D-> E-> F-> G | Treatment C-> B-> A-> J-> K-> L-> M-> N-> B | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (18.01) | 34.3 (7.51) | 42.3 (7.02) | 42.0 (6.32) | 34.7 (5.86) | 43.3 (8.50) | 38.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 0 | 2 | 5
  Male | 3 | 3 | 2 | 2 | 3 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 0 | 1 | 1 | 6
  Not Hispanic or Latino | 2 | 0 | 3 | 4 | 2 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 1 | 1 | 8
  White | 2 | 1 | 0 | 2 | 2 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCinf of Abrocitinib Following the Administration of Abrocitinib Commercial Tablet, Abrocitinib Oral Suspension Formulation 1 or Famotidine Plus Abrocitinib Commerical Tablet
Description: Area under the plasma concentration time profile from time 0 extrapolated to infinity (AUCinf) was measured. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Abrocitinib 200 mg Commercial Tablet: Abrocitinib 200 mg commercial tablet was administered on Day 1 under fasted conditions.
- Abrocitinib 200 mg Oral Suspension Formulation 1: Abrocitinib 200 mg oral suspension formulation 1 was administered on Day 1 under fasted conditions.
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet: Famotidine 40 mg tablet was administered 2 hours prior to abrocitinib 200 mg commercial tablet on Day 1 under fasted conditions.
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 18 | 18 | 18
nanogram*hour per milliliter (ng*hr/mL) | 4623 (66) | 4601 (54) | 3096 (61)
Statistical Analysis 1: Comparison: Abrocitinib 200 mg Commercial Tablet vs Abrocitinib 200 mg Oral Suspension Formulation 1; Test: Abrocitinib 200 mg oral suspension formulation 1; Reference: Abrocitinib 200 mg commercial tablet; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of adjusted geometric means = 96.96, 90% CI 2-sided [85.43 to 110.03]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg Commercial Tablet vs Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet; Test: Famotidine 40 mg tablet + Abrocitinib 200 mg commecial tablet; Reference: Abrocitinib 200 mg commercial tablet; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Ratio (%) of adjusted geometric means = 62.87, 90% CI 2-sided [54.85 to 72.07]

2. Primary Outcome: Cmax of Abrocitinib Following the Administration of Abrocitinib Commercial Tablet, Abrocitinib Oral Suspension Formulation 1 or Famotidine Plus Abrocitinib Commerical Tablet
Description: Maximum observed plasma concentration (Cmax) was measured. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 18 | 18 | 18
nanogram per milliliter (ng/mL) | 1264 (67) | 1218 (56) | 189.1 (77)
Statistical Analysis 1: Comparison: Abrocitinib 200 mg Commercial Tablet vs Abrocitinib 200 mg Oral Suspension Formulation 1; Test: Abrocitinib 200 mg oral suspension formulation 1; Reference: Abrocitinib 200 mg commercial tablet; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of adjusted geometric means = 100.07, 90% CI 2-sided [80.28 to 124.74]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg Commercial Tablet vs Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet; Test: Famotidine 40 mg tablet + Abrocitinib 200 mg commercial tablet; Reference: Abrocitinib 200 mg commercial tablet; Test type: Other — The ratio and 90% CI were expressed as percentages; Ratio (%) of adjusted geometric means = 15.53, 90% CI 2-sided [12.46 to 19.36]

3. Primary Outcome: Assessment of Overall Liking After Administering Each Abrocitinib Oral Suspension Formulation (Formulation [F]1-F6) in Part B
Description: For the taste assessment in Part B of the study, the data used in the analysis was transcribed and rescaled to a score from 0 to 100 from the raw measurements on the Taste Assessment Questionnaire. The score of 0 was considered Favorable and the score of 100 was considered Not Favorable. Higher score means more unfavorable.
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: All participants who had tasted the abrocitinib suspension formulations and made scores on the taste questionnaires were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Abrocitinib 200 mg Oral Suspension Formulation 1: Participants were given abrocitinib 200 mg oral suspension formulation 1.
- Abrocitinib 200 mg Oral Suspension Formulation 2: Participants were given abrocitinib 200 mg oral suspension formulation 2.
- Abrocitinib 200 mg Oral Suspension Formulation 3: Participants were given abrocitinib 200 mg oral suspension formulation 3.
- Abrocitinib 200 mg Oral Suspension Formulation 4: Participants were given abrocitinib 200 mg oral suspension formulation 4.
- Abrocitinib 200 mg Oral Suspension Formulation 5: Participants were given abrocitinib 200 mg oral suspension formulation 5.
- Abrocitinib 200 mg Oral Suspension Formulation 6: Participants were given abrocitinib 200 mg oral suspension formulation 6.
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 42.32 (35.117) | 72.10 (24.243) | 44.95 (34.422) | 42.19 (34.366) | 71.08 (27.491) | 69.29 (27.565)
  5 min | 40.21 (35.480) | 69.59 (25.882) | 42.83 (34.549) | 40.32 (32.691) | 71.87 (24.190) | 67.34 (27.632)
  10 min | 37.78 (34.025) | 65.65 (26.857) | 38.86 (30.808) | 33.90 (29.544) | 67.78 (24.919) | 62.89 (30.153)
  20 min | 35.55 (33.379) | 64.48 (27.644) | 37.56 (29.758) | 31.97 (29.563) | 61.68 (28.681) | 57.95 (28.483)

4. Primary Outcome: Assessment of Mouth Feel After Administering Each Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 40.12 (28.336) | 61.59 (26.218) | 40.79 (33.908) | 42.10 (30.178) | 63.59 (25.544) | 61.59 (31.543)
  5 min | 37.26 (27.903) | 54.22 (26.738) | 37.81 (33.045) | 38.67 (27.688) | 61.21 (25.335) | 60.48 (30.987)
  10 min | 35.61 (29.456) | 50.57 (26.578) | 35.18 (33.222) | 31.90 (24.808) | 55.33 (27.451) | 52.36 (31.626)
  20 min | 34.95 (30.347) | 42.22 (30.676) | 34.83 (33.221) | 26.89 (23.277) | 49.27 (29.356) | 44.33 (32.906)

5. Primary Outcome: Assessment of Bitterness After Administering Each Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 39.25 (30.773) | 64.25 (27.312) | 32.06 (27.383) | 28.63 (21.634) | 70.76 (27.869) | 63.28 (23.400)
  5 min | 36.54 (32.008) | 53.30 (30.392) | 31.14 (27.875) | 25.21 (19.685) | 63.62 (26.141) | 57.77 (28.066)
  10 min | 33.80 (31.609) | 47.72 (31.067) | 27.27 (25.124) | 20.95 (19.000) | 53.65 (25.657) | 49.41 (26.827)
  20 min | 30.83 (31.598) | 39.24 (31.325) | 24.92 (23.048) | 18.19 (19.554) | 45.56 (30.635) | 42.37 (27.755)

6. Primary Outcome: Assessment of Tongue/Mouth Burn After Administering Each Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 28.90 (26.489) | 41.87 (30.238) | 25.87 (23.920) | 26.89 (25.884) | 35.75 (30.848) | 41.05 (32.462)
  5 min | 24.48 (25.226) | 35.40 (28.451) | 22.86 (22.477) | 22.67 (24.999) | 28.76 (25.809) | 37.89 (33.134)
  10 min | 23.73 (26.631) | 31.24 (26.305) | 18.29 (20.001) | 18.29 (22.999) | 22.82 (25.042) | 36.99 (32.737)
  20 min | 21.65 (28.937) | 23.97 (26.386) | 15.40 (20.156) | 16.51 (22.374) | 17.68 (21.927) | 33.68 (32.903)

7. Primary Outcome: Assessment of Salty Taste After Administering Each Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 19.73 (26.872) | 39.52 (31.190) | 19.84 (21.560) | 21.84 (21.319) | 39.24 (30.962) | 34.98 (31.103)
  5 min | 19.34 (27.435) | 35.56 (28.372) | 13.78 (17.276) | 19.49 (22.504) | 33.43 (24.688) | 30.92 (30.413)
  10 min | 19.43 (27.776) | 29.49 (26.602) | 12.29 (17.121) | 15.94 (21.414) | 25.33 (22.853) | 31.85 (33.229)
  20 min | 19.61 (27.872) | 25.62 (26.613) | 12.35 (17.234) | 15.68 (21.290) | 20.89 (19.444) | 28.60 (28.337)

8. Primary Outcome: Assessment of Sour Taste After Administering Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 25.44 (26.343) | 52.54 (27.703) | 24.86 (24.663) | 25.65 (22.452) | 48.35 (34.210) | 47.37 (33.103)
  5 min | 24.54 (26.919) | 46.32 (28.172) | 21.75 (23.849) | 21.71 (22.198) | 41.02 (31.652) | 39.73 (32.655)
  10 min | 23.16 (27.074) | 42.44 (29.892) | 18.70 (21.879) | 19.18 (20.652) | 33.30 (31.797) | 36.33 (32.522)
  20 min | 21.68 (27.373) | 37.05 (30.426) | 16.95 (21.472) | 18.16 (20.241) | 28.98 (31.338) | 34.31 (31.151)

9. Primary Outcome: Assessment of Sweet Taste After Administering Abrocitinib Oral Suspension Formulation (F1-F6) in Part B
Description: as for outcome 3
Time Frame: 0 Hours, 5, 10, 20 min after swallowing the suspension on Day 1 of each period.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg Oral Suspension Formulation 1 | Abrocitinib 200 mg Oral Suspension Formulation 2 | Abrocitinib 200 mg Oral Suspension Formulation 3 | Abrocitinib 200 mg Oral Suspension Formulation 4 | Abrocitinib 200 mg Oral Suspension Formulation 5 | Abrocitinib 200 mg Oral Suspension Formulation 6
Number analyzed (Participants) | 19 | 18 | 18 | 18 | 18 | 19
Units on a scale
  0 Hours | 31.16 (26.157) | 82.16 (19.816) | 30.16 (29.536) | 27.90 (24.626) | 78.48 (28.017) | 74.53 (29.874)
  5 min | 38.02 (30.485) | 78.32 (23.269) | 33.14 (28.948) | 31.56 (29.205) | 76.60 (28.824) | 72.84 (29.862)
  10 min | 40.42 (32.265) | 78.35 (23.383) | 33.52 (29.713) | 32.38 (32.348) | 74.86 (29.812) | 64.81 (33.275)
  20 min | 44.54 (34.296) | 75.18 (26.743) | 35.46 (29.622) | 33.33 (31.472) | 73.46 (31.151) | 62.50 (33.720)

10. Secondary Outcome: AUCinf of Abrocitinib Metabolite (PF-06471658/M1) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Area under the plasma concentration time profile from time 0 extrapolated to infinity.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: The analysis population refers to all participants dosed who had at least 1 of the PK parameters of secondary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Abrocitinib 200 mg Commercial Tablet: Abrocitinib 200 mg commercial tablet was administered on Day 1, under fasted conditions.
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet: Famotidine 40 mg tablet was administered 2 hours prior to abrocitinib 200 mg commercial tablet under fasted conditions on Day 1.
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 18 | 13
ng*hr/mL | 1048 (34) | 903.2 (32)

11. Secondary Outcome: AUCinf of Abrocitinib Metabolite (PF-07055087/M2) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Area under the plasma concentration time profile from time 0 extrapolated to infinity.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 17 | 7
ng*hr/mL | 1369 (22) | 1108 (15)

12. Secondary Outcome: AUCinf of Abrocitinib Metabolite (PF-07054874/M4) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Area under the plasma concentration time profile from time 0 extrapolated to infinity.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 15 | 13
ng*hr/mL | 2139 (34) | 1705 (33)

13. Secondary Outcome: Cmax of Abrocitinib Metabolite (PF-06471658/M1) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 18 | 18
ng/mL | 216.8 (82) | 57.38 (55)

14. Secondary Outcome: Cmax of Abrocitinib Metabolite (PF-07055087/M2) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 18 | 18
ng/mL | 214.3 (58) | 56.42 (42)

15. Secondary Outcome: Cmax of Abrocitinib Metabolite (PF-07054874/M4) Following the Administration of Abrocitinib 1×200 mg Tablet With or Without Famotidine 40 mg in Part A
Description: Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose on Day 1 of each period.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet
Number analyzed (Participants) | 17 | 18
ng/mL | 400.5 (39) | 87.96 (47)

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Event
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product, without regard to relatedness. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Treatment-related TEAEs were any untoward medical occurrence attributed to study intervention. Relatedness to study intervention was determined by the investigator.
Time Frame: Baseline up to follow-up (Day 36)
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Abrocitinib 200 mg Commercial Tablet: In part A of the study, abrocitinib 200 mg commercial tablet was administered on Day 1 under fasted conditions.
- Abrocitinib 200 mg Oral Suspension Formulation 1: In part A of the study, abrocitinib 200 mg oral suspension formulation 1 was administered on Day 1 under fasted conditions.
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet: In part A of the study, famotidine 40 mg tablet + abrocitinib 200 mg commercial tablet were administered on Day 1 under fasted conditions.
- Abrocitinib 200 mg Oral Suspension Formulation 1-6: In part B of the study, abrocitinib 200 mg oral suspension formulation 1-6 were administered on Day 1 of each period under fasted conditions.
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6: In part B of the study, famotidine 40 mg tablet + abrocitinib 200 mg oral suspension formulation 1-6 were administered on Day 1 of each period under fasted conditions.
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1-6 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6
Number analyzed (Participants) | 18 | 18 | 18 | 9 | 10
Participants
  All-causality AEs | 6 | 8 | 6 | 5 | 2
  Treatment-related AEs | 3 | 5 | 0 | 4 | 0
  SAEs | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Participants with laboratory abnormalities (without regard to baseline abnormality) were reported.
Time Frame: Baseline up to follow-up (Day 36)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1-6 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6
Number analyzed (Participants) | 18 | 18 | 18 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Values
Description: Participants with clinically significant vital sign values were reported.
Time Frame: Baseline up to follow-up (Day 36)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1-6 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6
Number analyzed (Participants) | 18 | 18 | 18 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Values
Description: Participants with clinically significant abnormal ECG values were reported.
Time Frame: Baseline up to follow-up (Day 36)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1-6 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6
Number analyzed (Participants) | 18 | 18 | 18 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Nausea AEs
Description: Number of participants who received abrocitinib 200 mg alone and who received abrocitinib 200 mg plus famotidine 40 mg and had nausea AEs were reported.
Time Frame: Baseline up to follow-up (Day 36)
Population: All participants who received at least 1 dose of abrocitinib 200 mg alone or abrocitinib 200 mg plus famotidine 40 mg.
Measure: Count of Participants; unit: Participants
Groups:
- Abrocitinib 200 mg Alone: All participants in abrocitinib 200 mg commercial tablet and abrocitinib 200 mg oral suspension formulation 1 in Part A as well as sequence 4-6 in Part B were included.
- Abrocitinib 200 mg Plus Famotidine 40 mg: All participants in abrocitinib 200 mg commercial tablet plus famotidine 40 mg tablet in Part A as well as sequence 1-3 in Part B were included.
Arm/Group | Abrocitinib 200 mg Alone | Abrocitinib 200 mg Plus Famotidine 40 mg
Number analyzed (Participants) | 45 | 28
Participants | 12 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (Day 36)
Description: Occurrences of AEs in this study were reported according to the study interventions that participants received, according to the study safety objective. Abrocitinib 200 mg oral suspension formulations (with different flavors) were prepared with different levels of flavor and sweetener at study site, and any AEs occurrences for these study interventions were combined to ensure the presentation of safety profiles of Abrocitinib 200 mg oral suspension formulation.
Groups:
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet: In part A of the study, aamotidine 40 mg tablet + Abrocitinib 200 mg commercial tablet were administered on Day 1 under fasted conditions.
- Aborcitinib 200 mg Oral Suspension Formulation 1-6: In part B of the study, aborcitinib 200 mg oral suspension formulation 1-6 were administered on Day 1 od each period under fasting conditions.
- Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6: In part B of the study, famotidine 40 mg tablet + abrocitinib 200 mg oral suspension formulation 1-6 were administered on Day 1 of each period under fasting conditions.
Arm/Group | Abrocitinib 200 mg Commercial Tablet | Abrocitinib 200 mg Oral Suspension Formulation 1 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet | Aborcitinib 200 mg Oral Suspension Formulation 1-6 | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 6/18 | 8/18 | 6/18 | 5/9 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib 200 mg Commercial Tablet (N=18) | Abrocitinib 200 mg Oral Suspension Formulation 1 (N=18) | Famotidine 40 mg Tablet + Abrocitinib 200 mg Commercial Tablet (N=18) | Aborcitinib 200 mg Oral Suspension Formulation 1-6 (N=9) | Famotidine 40 mg Tablet + Abrocitinib 200 mg Oral Suspension Formulation 1-6 (N=10)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 0 | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 1 | 0
Hunger (General disorders) | 1 | 0 | 0 | 2 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04903093/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04903093/SAP_001.pdf